CLINICAL TRIAL: NCT05181384
Title: Pelvic Floor Muscles and Stabilization Integrated Training With Transabdominal Ultrasonography-guided Biofeedback Improved Pregnancy-related Pelvic Girdle Pain and Disability: A Randomized Controlled Trial
Brief Title: Pelvic Floor Muscles and Stabilization Integrated Training Improved Pregnancy-related Pelvic Girdle Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: YI-JU TSAI (Other)
Responsible Party: Sponsor-Investigator, YI-JU TSAI, professor, National Cheng Kung University
Organization: National Cheng Kung University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCKU_PPGP three group
Record Dates: First submitted 2021-11-24; First posted 2022-01-06 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Pelvic Girdle Pain
Keywords: Pregnancy-related pelvic girdle pain; Postpartum women; Pelvic stabilization exercise; Pelvic floor muscles; Ultrasonography imaging; Biofeedback
MeSH Terms: conditions — Pelvic Girdle Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Transabdominal Sonography-guided Biofeedback group (Experimental): pelvic floor muscle training with transabdominal sonography-guided Biofeedback
  Interventions: Other: isolated pelvic floor muscles training; Other: comprehensive stabilization exercise program; Other: education of pelvic girdle
- Exercise group (Active Comparator): pelvic floor muscle training
  Interventions: Other: isolated pelvic floor muscles training; Other: comprehensive stabilization exercise program; Other: education of pelvic girdle
- Control group (Placebo Comparator): pelvic girdle education
  Interventions: Other: education of pelvic girdle

INTERVENTIONS:
Other: isolated pelvic floor muscles training — isolated pelvic floor muscles training was emphasized, consisting of both quick and sustained contractions.
  Arms: Exercise group; Transabdominal Sonography-guided Biofeedback group
Other: comprehensive stabilization exercise program — incorporated the contraction of PFMs with other spinal or extremity muscles
  Arms: Exercise group; Transabdominal Sonography-guided Biofeedback group
Other: education of pelvic girdle — educational session includes pelvic anatomy, mechanism of and risk factors for PPGP, and proper posture or body mechanism

SUMMARY:
Pregnancy-related pelvic girdle pain (PPGP) is a common musculoskeletal problem for women during pregnancy and after delivery. The main purpose of this study was to investigate the effects of integrated training for pelvic floor muscles (PFMs) and stabilization with and without transabdominal ultrasonography (TAUS) imaging-guided biofeedback on pain, disability, and physical function, and muscle functions for the abdominal muscles and PFMs in postpartum women with PPGP.

DETAILED DESCRIPTION:
Many women have pregnancy-related pelvic girdle pain (PPGP), and about 30% with PPGP women still complain of pain after 1-year postpartum. Both physical and mental functions of PPGP women are impaired. Pelvic stabilization exercise with pelvic floor muscle training is believed to be effective for reducing pain and improved pelvic stability. However, intervention studies on PPGP women is limited and current evidence are controversial. Incorrect pelvic floor muscle activations may be partly contributed to these results. One previous study has showed about 60% of women cannot activate pelvic floor muscles correctly. Transabdominal sonography-guided biofeedback by observing bladder movements is no-invasive and benefit learning correct muscle contraction. Therefore, the main purposes for this study are to investigate the effects of pelvic stabilization training using transabdominal sonography-guided biofeedback in postpartum women with PPGP. A total of 50 postpartum PPGP women will be randomized into one of the two groups: (1) biofeedback group, (2) exercise group, (3) control group, and (4) health group. Subjects in the biofeedback group and exercise group will perform the same exercise training for 8 weeks except the subjects in the biofeedback group will receive transabdominal sonography-guided biofeedback of bladder movement for the first 4 weeks. The outcome assessment will include the muscle thickness of abdominal muscle and pelvic floor muscle control, functional performance of ASLR fatigue task, timed up and go and fast walking, pelvic girdle questionnaire (PGQ), and numeric rating scale (NRS). It is anticipated that the biofeedback group will have more improvements that the exercise group.

ELIGIBILITY:
Inclusion Criteria:

* postpartum : ≥ 3 months
* pregnancy-related pelvic pain
* pain location is located between posterior iliac crest and gluteal fold
* Clinical screening test for pelvic pain: ASLR : positive and SI joint ≥ 2 (+ symphysis ≥ 1)

Exclusion Criteria:

* lumbar or pelvic surgery
* lother causes of pelvic pain (such as fractures)
* lRadiculopathy
* lother health problems, such as cancer, cardiovascular disease, rheumatism , etc
* ldaily activities limited , unable to complete the experiment
* lcommunication disorders
* lmental disorder
* lpregnancy
* lhave been trained in stable muscle strength in the past.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
pain intensity measure of Numeric Rating Scale (NRS) | Change from baseline to 8 weeks
  Numeric Rating Scale (NRS) is a self-reported instrument assessing average pain intensity in currently. Possible score range from 0 (no pain) to 10 (worst possible pain).
pain intensity measure of pelvic girdle questionnaire(PGQ) | Change from baseline to 8 weeks
  pelvic girdle questionnaire(PGQ) is a self-reported instrument assessing pelvic girdle pain intensity in currently. Questionnaire consisting of 20 activity items and 5 symptom items on a 4-point response scale. Possible score range from 0 (no pain) to 100 (worst possible pain).

SECONDARY OUTCOMES:
functional performance of ASLR fatigue task | Change from baseline to 8 weeks
  Participants lifted the heel of the test leg to 20 cm for as long as possible. Participants were required to maintain pressure in the cuff beneath their back as close to 40 mm Hg as possible. Visual feedback of cuff pressure was provided throughout the task, but no instruction was given on how to affect cuff pressure. Task failure was defi ned as an inability to maintain heel height 10 cm or more off the plinth and/or a change in cuff pressure of 20 mm Hg or more.
functional performance of timed up and go test | Change from baseline to 8 weeks
  Test instructions were given in Norwegian. Translated into English, the instructions were as follows: 'After "ready, set, go" stand up, walk as fast as you can until you cross the white line, turn around, and walk back to the chair and sit down again'. The white line was positioned 3m from the patient's starting position.
  'After "ready, set, go" stand up, walk as fast as you can until you cross the white line, turn around, and walk back to the chair and sit down again'. The white line was positioned 3m from the patient's starting position.
functional performance of 6m timed walk test (fast walking) | Change from baseline to 8 weeks
  Subjects commenced the test in standing with their toes up against the tape marker. Test instructions translated into English were as follows: 'After "ready, set, go", walk as fast as you can up to the last white line without stopping or speaking along the way'. Performances were timed (to the nearest 100th of a second) between the 2m and 8m markers and later converted into speed in metres per second.
Muscle function measures of abdominal muscle | Change from baseline to 8 weeks
  Untrasonography image for muscle thickness of abdominal muscle during rest and ASLR test.
Muscle function measures of pelvic floor muscle control | Change from baseline to 8 weeks
  Untrasonography image for muscle thickness of pelvic floor muscle control at maximum contraction.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University, Tainan, Taiwan